CLINICAL TRIAL: NCT02772302
Title: Feasibility Study of the mindBEAGLE Device in Patients With Disorders of Consciousness or Locked-In Syndrome
Brief Title: Feasibility of mindBEAGLE in Disorders of Consciousness or Locked-In Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Brian L. Edlow, M.D., Instructor of Neurology, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2015P002731
Record Dates: First submitted 2016-03-30; First posted 2016-05-13 (Estimated); Results first posted 2021-04-30 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-06

CONDITIONS: Consciousness Disorders; Locked-In Syndrome
MeSH Terms: conditions — Consciousness Disorders; Locked-In Syndrome

STUDY DESIGN:
Intervention Model Description: Arm 1: patients Arm 2: healthy controls
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients (Experimental): Application of bedside, EEG-based mindBEAGLE Brain-Computer Interface
  Interventions: Device: mindBEAGLE EEG-based brain-computer interface
- Healthy Controls (Experimental): Application of bedside, EEG-based mindBEAGLE Brain-Computer Interface
  Interventions: Device: mindBEAGLE EEG-based brain-computer interface

INTERVENTIONS:
Device: mindBEAGLE EEG-based brain-computer interface

SUMMARY:
The primary aims of this study are:

1. To determine the feasibility of deploying mindBEAGLE, a portable, bedside EEG-based system, in the Intensive Care Unit in patients with disorders of consciousness (DOC) or locked-in syndrome (LIS);
2. To determine if mindBEAGLE neurophysiologic markers of cognitive function correlate with bedside behavioral assessments of consciousness;
3. To determine if mindBEAGLE neurophysiologic markers of cognitive function correlate with functional MRI (fMRI) and electroencephalography (EEG) biomarkers of consciousness;
4. To determine if mindBEAGLE can serve as an assistive communication device for people with LIS.

DETAILED DESCRIPTION:
1. To determine the feasibility of deploying mindBEAGLE, a portable, bedside EEG-based system, in the Neurosciences Intensive Care Unit in patients with DOC or LIS;
2. To determine if mindBEAGLE neurophysiologic markers of cognitive function correlate with bedside behavioral assessments of consciousness;
3. To determine if mindBEAGLE can serve as an assistive communication device for people with LIS.

ELIGIBILITY:
Inclusion Criteria:

* Age>18
* Diagnosis of coma
* Vegetative state
* Minimally conscious state
* Confusional state
* Locked-in state

Exclusion Criteria:

• History of developmental, neurologic, or major psychiatric disorder resulting in functional disability

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian L. Edlow, M.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- See also: Feasibility of an EEG-based brain-computer interface in the intensive care unit — https://pubmed.ncbi.nlm.nih.gov/29804044/

RESULTS

PARTICIPANT FLOW:
Groups:
- mindBEAGLE: Application of bedside, EEG-based mindBEAGLE Brain-Computer Interface
  mindBEAGLE EEG-based brain-computer interface
- Healthy Controls: healthy subjects with no history of neurological disease
Period: Overall Study
Arm/Group | mindBEAGLE | Healthy Controls
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- mindBEAGLE (Inpatient Participants): Application of bedside, EEG-based mindBEAGLE Brain-Computer Interface
  mindBEAGLE EEG-based brain-computer interface
- mindBEAGLE (Healthy Controls): Application of bedside, EEG-based mindBEAGLE Brain-Computer Interface tested in healthy controls to provide baseline validation of the technology.
- Total: Total of all reporting groups
Arm/Group | mindBEAGLE (Inpatient Participants) | mindBEAGLE (Healthy Controls) | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 3 | 1 | 4
Age, Continuous [Median (Full Range); unit: years] | 56 [37 to 72] | 34 [20 to 70] | 41 [20 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 8 | 6 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 5 | 9
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 20

OUTCOME MEASURES:

1. Primary Outcome: Behavioral Diagnosis of Level of Consciousness (LoC)
Description: LoC will be defined using the Coma Recovery Scale-Revised behavioral evaluation (score range 0-23). Higher scores are generally associated with a higher level of consciousness.
Time Frame: on the day of intervention
Population: patients in the ICU (n=10) and healthy control subjects (n=10)
Measure: Number; unit: score on a scale
Groups:
- Healthy Control Subjects: Application of bedside, EEG-based mindBEAGLE Brain-Computer Interface mindBEAGLE EEG-based brain-computer interface
Arm/Group | mindBEAGLE | Healthy Control Subjects
Number analyzed (Participants) | 10 | 10
score on a scale
  patient 1 | 0 | 23
  patient 2 | 2 | 23
  patient 3 | 2 | 23
  patient 4 | 2 | 23
  patient 5 | 5 | 23
  patient 6 | 3 | 23
  patient 7 | 10 | 23
  patient 8 | 13 | 23
  patient 9 | 16 | 23
  patient 10 | 16 | 23

ADVERSE EVENTS:
Time Frame: During mindBEAGLE assessment in the intensive care unit, which lasted up to 4 hours.
Description: Participants with Disorders of Consciousness or Locked in Syndrome were enrolled in the Neuro-ICU where adverse events, related or unrelated to the intervention/device were systematically monitored through regular investigator assessment and regular laboratory testing.
Arm/Group | mindBEAGLE | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | mindBEAGLE (N=10) | Healthy Controls (N=10)
Hypotension (General disorders) | 1 | NA — One serious, unexpected and unrelated adverse event was experienced, related to hypotension requiring IV fluid administration during EEG.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT02772302/Prot_SAP_000.pdf